Title: Comparison of traditional back-loaded fiducial needles with preloaded fiducial needles in EUS-guided fiducial marker placement for image-guided radiation therapy in patients with pancreatic cancer: A multicenter randomized controlled trial.

NCT02332863

Date: 11/27/2019

## Statistical Analysis Plan

The sample-size calculation was based on limited experimental data in a porcine model, and on a consensus decision among expert endosonographers regarding the relative reduction in the time (60%) to deploy preloaded fiducial markers<sup>18</sup>. We estimated that a sample size of 40 patients (20 in each arm) was needed to provide the study with at least 80% power and a 2-sided alpha of 0.05. All analyses were performed according to the intention-to-treat principle. Per-protocol analysis was also performed. Descriptive statistics are reported as absolute values (percentage), mean 2 standard deviation, and median (IQR), as appropriate. Comparisons of baseline characteristics and outcomes were evaluated using chi-square or Fischer exact test for categorical data and Student t test or Mann-Whitney U test for continuous data. Pre-established subgroup analysis was performed by tumor location (head/neck vs body/tail). Although not pre-established in the study protocol, results were also stratified by time of randomization (first half vs second half) to explore a possible learning curve effect. Statistical significance was defined as P <.05. All statistical analyses were performed using Stata/ IC version 12.1 (College Station, TX).

## References:

18. Draganov P.V., Chavalitdhamrong D., and Wagh M.S.: Evaluation of a new endoscopic ultrasound-guided multi-fiducial delivery system: a prospective non-survival study in a live porcine model. Dig Endosc 2013; 25: pp. 615-621